CLINICAL TRIAL: NCT01960582
Title: Housing Adaptations and Mobility Devices - Evaluation of a New Practice Strategy
Brief Title: Evaluation of Housing Adaptations and Mobility Devices
Acronym: FORMASEvid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Agneta Malmgren Fänge, Associate professor, Lund University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FORMAS 2011-907
Record Dates: First submitted 2013-09-27; First posted 2013-10-10 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Activities of Daily Living; Cost Effectiveness; Housing
Keywords: Housing adaptation; Independence; Costs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- New Practice Strategy (Experimental): Structured strategy for assessment and evaluation before and after intervention
  Interventions: Behavioral: New Practice Strategy
- Ordinary practice (No Intervention): Ordinary practice, not structured

INTERVENTIONS:
Behavioral: New Practice Strategy — Application of a structured case management strategy on housing adaptation cases
  Arms: New Practice Strategy

SUMMARY:
The rationale underlying this project is the fact that HA is a very common compensatory interven¬tion within municipality health care, undertaken to support an independent living in the own home. In addition, MD are frequently prescribed and used among HA clients in order to compensate for declined body functions. In spite of this, knowledge of their effects for the individual and the society is still scarce. In particular, systematic, evidence-based strategies based on clear-cut conceptual definitions and descriptions of procedures are lacking. Such strategies are crucial in order to evaluate the effects of HA and MD. In addition, longterm cost-effectiveness evaluations are crucial for policy implementation.

The overarching aim is to investigate outcomes of HA on aspects of home and health for sub-groups of persons with disabilities.

The specific aims are to:

* Investigate the effects of HA on home and health related outcomes, i.e. usability, fear of falling, activity/participation and health-related quality of life for different subgroups of persons, e.g. MD users and non MD-users
* Investigate the use of a new practice strategy for HA on home and health related outcomes for subgroups of persons with disabilities in terms of differences between municipalities
* Investigate societal level outcomes of HA and MD, i.e. costs and quality adjusted life years
* Gain a deeper understanding of the processes behind changes in outcomes We hypothesise that using a structure strategy for housing adaptation and mobility devices case management in ordinary practice in Swedish municipalities increase activity, participation, the usability of the home, and reduces societal costs.

DETAILED DESCRIPTION:
The ultimate goal of the project is to improve the housing situation of older people and people with disabilities, by determining the long term effects of housing adaptations (HA) for clients and society, and transferring this knowledge into guidelines for practitioners in the housing and building planning sector.

Specific research questions are:

RQ1. What are the long-term effects of HA for clients (individual goals achievement, activity, participation, health-related quality of life, usability, falls, functional capacity and use of mobility devices (MD), mortality, health care and social services consumption, and relocation)? RQ2. What are the long-term effects of HA for society (costs and cost- effectiveness)? RQ3. What are the barriers and facilitators to knowledge transfer in the area of HA? RQ4. How can evidence based knowledge be transferred into practical guidelines for housing and building planning in Sweden?

ELIGIBILITY:
Inclusion Criteria:

* Persons receiving housing adaptation
* Above 20 years

Exclusion Criteria:

* Persons with language deficits and/or cognitive decline

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2013-01-11 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
ADL Staircase | Differences in changes between intervention and control sites at baseline and 3, 6,12, 24 and 36 months after
  The ADL Staircase measures dependence on other persons in daily activities. Combined interview and observation

SECONDARY OUTCOMES:
Falls Efficacy Scale- FES-I | Differences in changes between intervention and control sites at baseline and 3, 6, 12, 24 and 36 months after
  FES-I measures perceived fear of falling

OTHER OUTCOMES:
Usability of the home, UIMH | Differences in changes between intervention and control sites between baseline and 3, 6,12,24 and 36 months after
  Self-rated assessment measuring the extent to which the person can perform Daily activities in the housing
Costs of housing adaptations | 3,6, 12, 24 and 36 months after, for the whole sample
  The actual costs for the housing adaptation, including costs for travel, work hours, and material will be calculated based on invoices benefit
Cost-benefit for client and society | At 24 and 36 months after the housing adaptation, for the whole sample
  The cost-benefit of the housing adaptation will be calculated based on health economic models utilising data from EQ-5D instrument

CONTACTS AND LOCATIONS:
Overall Officials: Agneta M Fänge, PhD, Principal Investigator — Lund University
Locations (1):
- Department of Health Sciences, Lund University, Lund, Sweden

REFERENCES:
- [Derived] Malmgren Fange A, Carlsson G, Axmon A, Thordardottir B, Chiatti C, Nilsson MH, Ekstam L. Effects of applying a standardized assessment and evaluation protocol in housing adaptation implementation - results from a quasi-experimental study. BMC Public Health. 2019 Nov 4;19(1):1446. doi: 10.1186/s12889-019-7815-9. PMID 31684916
- [Derived] Ekstam L, Carlsson G, Chiatti C, Nilsson MH, Malmgren Fange A. A research-based strategy for managing housing adaptations: study protocol for a quasi-experimental trial. BMC Health Serv Res. 2014 Nov 29;14:602. doi: 10.1186/s12913-014-0602-5. PMID 25432718